CLINICAL TRIAL: NCT00448253
Title: Safety and Pharmacokinetics of Anthrax Immune Globulin Intravenous (Human), NP-015, in Healthy Volunteers.
Brief Title: Safety and Pharmacokinetic Study of Anthrax Immune Globulin Derived From Human Serum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AX001
Record Dates: First submitted 2007-03-14; First posted 2007-03-16 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Symptoms of Inhalational Anthrax
Keywords: Inhalational Anthrax; Human Immune globulin
MeSH Terms: conditions — Inhalation anthrax | interventions — Anthrax Immune Globulin Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Three Cohorts evaluating three dosage levels: 210, 420 or 840 units TNA. And a Fourth Cohort at 840 units TNA with 2 additional product lots.
  Interventions: Biological: NP-015
- 2 (Placebo Comparator): Saline (equal volume to 210 U, 420 U, or 840 U TNA dose)
  Interventions: Biological: NP-015

INTERVENTIONS:
Biological: NP-015 — Three Cohorts evaluating three dosage levels: 210, 420 or 840 units TNA, or placebo.
  And a Fourth Cohort at 840 units TNA with 2 additional product lots.
  Other Names: Anthrax Immune Globulin (AIG)

SUMMARY:
The purpose of the study is to assess the pharmacokinetics of three doses of NP-015 (210, 420 or 840 units TNA) in healthy volunteers. To evaluate the safety of NP-015 based on adverse events and laboratory assessments. To determine the dose proportionality relation of three different doses of NP-015.

DETAILED DESCRIPTION:
* The test product is Anthrax Immune Globulin Intravenous (Human), NP-015.
* The product is supplied as a sterile liquid suitable for IV administration.
* Product potency is expressed in units of anthrax toxin neutralization assays(TNA) per vial.
* This study is a phase 1, placebo controlled, dose-ranging study in healthy volunteers. Subjects will receive one of three NP-015 doses (210, 420 or 840 units TNA) or equal volumes of saline placebo.
* Enrolment will be sequential, starting at the lowest NP-015 dose with accrual into the next higher dose after all patients at the lower dose have been treated.
* The first 3 Cohorts: The Subjects will be recruited in cohorts of 24, with placebo controls included in each dosing group. In each cohort, subjects will be randomized to receive either NP-015 (N = 18/dosing group) or placebo (N = 6/dosing group). For Cohort 4: 20 Subjects will be recruited and dosed at the highest dose with 2 additional product lots (10 subjects per lot).

Plasma samples will be drawn over 84 days. Plasma will be tested for anti-anthrax antibodies by a protective antigen (anti-PA) ELISA and toxin neutralization assay (TNA).

* Serological testing for HIV, HBV and HCV will be conducted at screening to determine eligibility. Nucleic acid amplification testing (NAT) and serological testing for HIV, HBV and HCV will be conducted at baseline (day -1) and at the final visit (day 84 or early withdrawal). NAT for parvovirus B19 will be conducted at baseline (day -1), day 14, and the final visit (day 84 or early withdrawal).
* Safety data will be collected throughout the 84-day study.

Screening (within 28 days prior to Baseline):

* Informed consent
* Review of admission criteria
* Medical history, general physical examination, vital signs, electrocardiogram and concomitant medications will be recorded
* Hematology, blood chemistry, urinalysis, viral serology (anti-HIV-1/2, Anti-HCV, HBsAg, anti-HBc)
* Serum pregnancy test for all female subjects
* Drug screen (urine)
* Blood collection for anti-PA antibody and toxin neutralization assay (TNA) assessment

Baseline (Day -1, within 24 hours prior to Day 0)

* Review of admission criteria
* Assessment of brief physical exam, vital signs, weight, hematology, blood chemistry, urinalysis, and concomitant medications
* Assessment of haptoglobin and free hemoglobin levels
* Update of medical history
* NAT testing for HIV, HBV, HCV and parvovirus B19, and serological testing for HIV, HBV and HCV
* Serum pregnancy test for all female subjects
* Alcohol (urine) and drug screen (urine)
* Blood collection for baseline anti-PA antibody and TNA assessment
* Subjects will be required to stay overnight following their baseline assessment

NP-015 Administration (day 0)

* Following baseline assessment, NP-015 will be administered intravenously
* Urinalysis will be performed at the end of the infusion period (appearance and color, specific gravity, protein, glucose, pH, occult blood, ketones, microscopic examination)

Assessments following the completion of NP-015 administration (1, 3 and 8 hrs; days 1, 3, 5, 7, 9, 11, 14, 21, 28, 42, 56 and 84 or early withdrawal)

* Following NP-015 administration, blood will be collected for anti-PA antibody ELISA analysis and TNA assessment at each of the respective times.
* Assessment of vital signs, adverse events and concomitant medications.

Additional Assessments:

* Days 1, 3, 7, 14, 28 and 84 or early withdrawal: Assessment of hematology, blood chemistry and urinalysis.
* Day 1: Assessment of haptoglobin and free hemoglobin levels.
* Day 14: NAT for parvovirus B19.
* Day 28: serum pregnancy test for female subjects.
* Final (day 84 or early withdrawal) visit: a general physical exam, serum pregnancy test for female subjects, and viral marker testing (NAT for HBV, HCV, HIV and parvovirus B19, and serology for HIV, HBV and HCV) will be performed.

For Cohort 4 there will be no anti anthrax antibody testing and the subjects will be assessed for safety only, up to day 28.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18/19 (dependent on local age of majority) - 55 years
* Body mass index of 19 - 29
* For female subjects that are not surgically sterilized, willingness to use an effective method of contraception throughout the trial including:
* Using hormonal contraception (oral, injectable or implant) continuously for 3 months prior to the start of the trial and willing to continue to use hormonal contraception throughout the entire trial.
* IUD inserted at least 3 months prior to dosing.
* For female subjects who are postmenopausal < 2 years an FSH ≥ 40 mIU/mL must be obtained. If the FSH is < 40 mIU/mL the subject must agree to use an acceptable form of contraception (see above).
* For males that have not had a vasectomy, willingness to use a condom with spermicide for the duration of the study. Also, male subjects must not donate sperm for the duration of the study.
* Normal and healthy as determined by medical history, physical exam, ECG, vital signs and laboratory tests of liver, kidney and hematological functions
* Written informed consent

Exclusion Criteria:

* Heavy smokers (>10 cigarettes/day) or individuals using smokeless tobacco or nicotine containing products
* Use of any investigational product within the past 30 days
* Recipient of any blood product within the past 12 months
* Plasma donation within 7 days or significant blood loss or blood donation within 56 days of baseline
* Females with a hemoglobin level < 12 g/dL
* Males with a hemoglobin level < 13 g/dL
* History of hypersensitivity to blood products
* History of allergy to latex or rubber
* History of IgA deficiency
* Pregnancy or lactation
* Positive serology test for HIV or HCV, positive test for HBV as determined by HBsAg.
* History of, or suspected substance abuse problem (including alcohol)
* Failure of drug test at screening or baseline
* Failure of alcohol test at baseline or consumption of alcoholic beverages within 48 hours of baseline
* History of anthrax vaccination with AVA or any other anthrax vaccine
* Individuals with planned medical procedures that will occur during the study
* Use of prescription medications within 7 days prior to baseline, or anticipated use during the study (with the exception of hormonal contraceptives for females)
* Use of over-the-counter, herbal medications or vitamins within 7 days of study admission
* An opinion of the investigator that it would be unwise to allow participation of the subject in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Anti-PA antibody and TNA for PK analyses. | screen, baseline, and D0 hours 1,3,8 and day(s) 1,3,5,7,9,11,14,21,28,42,56 and 84

SECONDARY OUTCOMES:
Viral Markers for safety. | screen, baseline, and Day(s)14 and 84
Dose proportionality analyses. | screen, baseline, and D0 hours 1,3,8 and day(s) 1,3,5,7,9,11,14,21,28,42,56 and 84
Blood Chemistry | screen, baseline, and D0 hours 0,1,2 and day(s) 1,3,7,14,28, and 84
Urinalysis | screen, baseline, and D0 hours 0 and day(s) 1,3,7,14,28, and 84
Hematology (haptoglobin and free hemoglobin at baseline and day 1) | screen, baseline, Day(s) 1,3,7,14,28, and 84

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Marion, MD, PhD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States